CLINICAL TRIAL: NCT02977455
Title: Study on the Neurovascular Coupling Function in Patients Undergoing Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 304460568
Record Dates: First submitted 2016-11-16; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-10

CONDITIONS: Neurovascular Coupling Mechanism and Cognitive Function

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

SUMMARY:
Existing researches show that brain is an organ highly dependent on continuous blood supply. Energy and oxygen required for normal physiological activities in the brain are stably maintained by a neurovascular regulatory mechanism, also known as functional congestion. While under pathological condition such as ischemia, this regulatory mechanism would be impaired and brain function loss and tissue damage occur. During anesthesia in cardiac surgery, inevitable circulatory fluctuations could result in decreasing blood pressure and cerebral blood flow and therefore brain tissue is in ischemia. In this situation the neurovascular regulatory mechanism will function and the brain oxygen saturation also changes based on how this mechanism is influenced. the investigators were devoted to observe how this mechanism was influenced during surgery and how the neural function recovers after surgery so to explore the relationship between them.

DETAILED DESCRIPTION:
Preoperative: Routine examinations, including pulse, blood pressure, electrocardiogram, hematological and biochemical tests from blood and urine. Anesthetist paid visit to patient and made judgement whether patient could be included or not based on rating of cognition. Anesthetist also introduced the research plan in detail and patient or guardian signed consent out of participants' own free will.

Intraoperative:

1. After admission, the investigators recorded regular vital signs and measured basic cerebral oxygen saturation, then inducted anesthesia.
2. After induction the investigators recorded anesthetic dose, vital signs and measured cerebral blood flow and oxygen saturation changes.
3. Using BIS to monitor we controlled the anesthesia depth at BIS value of 40 to 60.
4. Assuring patient's vital signs to be stable and safe, the investigators gave propofol (3 mg/kg, from Fresenius Kabi) intravenously when BIS was greater than 60 and observed while recorded any changes in BIS value, cerebral blood flow and oxygen saturation.

Postoperative: Patient was transferred to chest surgery ICU and vital signs were recorded.

Clinical data record:

General information: including name, gender, age, height, weight, education, name of disease, surgery method, admission number, ID number, address, contact information and so on;

Preoperative: cardiovascular medicine, vasoactive drugs, lab test results, result reviews, cognition rating and cerebral blood oxygen saturation basic value;

Intraoperative: circulatory parameters, medicine, temperature, BIS value, cerebral blood oxygen saturation and blood flow parameters;

Postoperative: extubation time, time of vasoactive drug administration, cognition rating (postoperative day 3 and day 7), postoperative complications (sudden cardiac death, disturbance of consciousness, pulmonary infection, acute lung injury, acute pulmonary embolism, cerebral infarction and so on);

Postoperative stay in hospital, ICU stay time, hospitalization cost, readmission, mortality (one, three and six months) and so on.

Cognition rating chart: based on "Direction of Chinese Binet Tests (third edition)".

ELIGIBILITY:
Inclusion Criteria:

1. Age <12 years old
2. Will take cardiac surgery and general anesthesia
3. Cognitive status is normal
4. Cardiac function grade Ⅱ-Ⅲ (using the NYHA cardiac function classification)

Exclusion Criteria:

1. Emergency surgery
2. ASA-V or VI
3. Coagulation disorders,multiple organs dysfunction, endocrine system diseases and severe infectious diseases
4. Patients have been installed pacemakers
5. Suspected or indeed alcohol, drug abuse history
6. Can not cooperate with research, such as the following: language understanding, mental illness, etc.
7. Participated in other clinical trials
8. Perioperative stroke
9. The researchers believe that should not be included in the study

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Cardiac surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Thirty of participants with Cognitive function assessment based on "Direction of Chinese Binet Tests (third edition)" | 6 months
  IQ scores will be used to quantify cognitive function